CLINICAL TRIAL: NCT02059044
Title: Information Systems-enabled Outreach Program for Adverse Drug Events
Acronym: ISTOP-ADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McGill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20130285; MOP125975 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2014-01-10; First posted 2014-02-11 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Adverse Drug Events
Keywords: patient safety; pharmacoepidemiology; health services research; adherence; information technology
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISTOP-ADE (Experimental): Interactive Voice Response System + Pharmacist
  Interventions: Other: ISTOP-ADE
- Routine care (No Intervention): Routine care

INTERVENTIONS:
Other: ISTOP-ADE — Interactive Voice Response System + Pharmacist
  Arms: ISTOP-ADE

SUMMARY:
One of the most common health care interventions in any healthcare setting is a medication prescription. Unfortunately, up to 25% of outpatient prescriptions are associated with adverse drug events (ADEs). ADEs decrease patient health directly and can lead to non-adherence, which in turn has negative consequences.

The investigators recently conducted a pilot project in which the feasibility and potential utility of an information technology enabled outreach program for monitoring patients receiving an outpatient prescription was tested. This intervention involved the use of an interactive voice response system programmed to automatically call ambulatory care patients following a prescription. If the system identified a potential medication problem, a pharmacist was notified who contacted the patient, modified the therapy accordingly, and informed a physician when necessary.

The pilot project included 568 patients with diverse illnesses in two Canadian cities. High levels of patient and provider acceptability of the system were determined from 21 day interviews. The program identified 56 of 125 (45%) ADEs and 10 of 26 (30%) of primary non-compliance events. Very few episodes of ameliorable ADEs were observed.

The investigators feel these results justify a randomized control trial to assess the effectiveness of the intervention for improving patient centered outcomes. Ambulatory care patients receiving incident prescriptions for one of four conditions (hypertension, diabetes mellitus, depression, and anxiety) will be randomized to the intervention or routine care. The investigators expect that the system will reduce the severity and duration of outpatient ADEs and improve adherence to medication care.

DETAILED DESCRIPTION:
One of the most common health care interventions in any healthcare setting is a medication prescription. On an individual and population level, outpatient medication use has the potential to improve health. Unfortunately, up to 25% of outpatient prescriptions are associated with adverse drug events (ADEs). ADEs decrease patient health directly and can lead to non-adherence, which in turn has negative consequences.

The investigators recently conducted a pilot project in which the feasibility and potential utility of an information technology enabled outreach program for monitoring patients receiving an outpatient prescription was tested. This intervention involved the use of an interactive voice response system programmed to automatically call ambulatory care patients following a prescription. If the system identified a potential medication problem, a pharmacist was notified who subsequently contacted the patient, modified the therapy accordingly, and informed a physician when necessary.

The pilot project included 568 patients with diverse illnesses in two Canadian cities (Montreal and Quebec City). The system successfully contacted 477 patients (84%). High levels of patient and provider acceptability of the system were determined from 21 day interviews. The program identified 56 of 125 (45%) ADEs and 10 of 26 (30%) of primary non compliance events. Very few episodes of ameliorable ADEs were observed in which the ADE severity could have been diminished with more appropriate management.

The investigators feel these results justify a randomized control trial to assess the effectiveness of our intervention for improving patient-centered outcomes. To determine whether the system reduces the severity and duration of outpatient ADEs and improves adherence to medication care at three and 12 months, ambulatory care patients receiving incident prescriptions for one of four conditions (hypertension, diabetes mellitus, depression, and anxiety) will be randomized to the intervention or routine care. As an exploratory analysis, the impact of the intervention on patient self efficacy and health services use will also be examined.

This study will help to define whether this promising intervention can improve patient health from both the individual patient and population health perspective. There is a wide scope of potential applications for this approach. This study will provide important information to guide these future applications beyond the specific question asked in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* spoken language is French or English
* physician is a user of MOXXI (electronic health record system) and patient has consented to be captured by MOXXI
* receiving a high-risk incident prescription
* medication insurance through Regie de l'Assurances Maladie du Quebec (RAMQ) insurance program

Exclusion Criteria:

* patient not appropriate for inclusion (as determined by prescribing physician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Failure to persist with medication regimen | 6 months

SECONDARY OUTCOMES:
Proportion of patients experiencing an ADE | within 30 days of prescription
Duration of symptoms attributable to the ADE from start to resolution | within 21 days following prescription
ADE resulting in an Emergency Department (ED) or inpatient encounter | within 21 days following prescription
ADE severity | within 30 days of prescription
Proportion of patients experiencing an ameliorable ADE | within 30 days of prescription
  An ameliorable ADE is an ADE whose severity should have been reduced if the healthcare system responded to the patient's health issues in an appropriate manner
Healthcare utilization (number of visits to MDs, EDs, days in hospital, and medication claims) | 1 year

OTHER OUTCOMES:
Cost of intervention for each patient | 21 days following prescription (average)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Forster, MD FRCPC MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oake N, Jennings A, van Walraven C, Forster AJ. Interactive voice response systems for improving delivery of ambulatory care. Am J Manag Care. 2009 Jun;15(6):383-91. PMID 19514804
- [Background] Forster AJ, Boyle L, Shojania KG, Feasby TE, van Walraven C. Identifying patients with post-discharge care problems using an interactive voice response system. J Gen Intern Med. 2009 Apr;24(4):520-5. doi: 10.1007/s11606-009-0910-3. Epub 2009 Jan 21. PMID 19156467
- [Background] Forster AJ, LaBranche R, McKim R, Faught JW, Feasby TE, Janes-Kelley S, Shojania KG, van Walraven C. Automated patient assessments after outpatient surgery using an interactive voice response system. Am J Manag Care. 2008 Jul;14(7):429-36. PMID 18611094
- [Background] Forster AJ, van Walraven C. Using an interactive voice response system to improve patient safety following hospital discharge. J Eval Clin Pract. 2007 Jun;13(3):346-51. doi: 10.1111/j.1365-2753.2006.00702.x. PMID 17518797
- [Background] Oake N, van Walraven C, Rodger MA, Forster AJ. Effect of an interactive voice response system on oral anticoagulant management. CMAJ. 2009 Apr 28;180(9):927-33. doi: 10.1503/cmaj.081659. PMID 19398739
- [Background] Auger C, Forster AJ, Oake N, Tamblyn R. Usability of a computerised drug monitoring programme to detect adverse drug events and non-compliance in outpatient ambulatory care. BMJ Qual Saf. 2013 Apr;22(4):306-16. doi: 10.1136/bmjqs-2012-001492. Epub 2013 Feb 8. PMID 23396853
- [Background] Forster AJ, Auger C; ISTOP ADE Investigators. Using information technology to improve the monitoring of outpatient prescribing. JAMA Intern Med. 2013 Mar 11;173(5):382-4. doi: 10.1001/jamainternmed.2013.2002. No abstract available. PMID 23381469
- [Derived] Forster AJ, Erlanger TE, Jennings A, Auger C, Buckeridge D, van Walraven C, Tamblyn R. Effectiveness of a computerized drug-monitoring program to detect and prevent adverse drug events and medication non-adherence in outpatient ambulatory care: study protocol of a randomized controlled trial. Trials. 2015 Jan 8;16:2. doi: 10.1186/1745-6215-16-2. PMID 25572800